CLINICAL TRIAL: NCT06576271
Title: A Phase 1, First-time-in-human, Three-part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of GSK4527363 in Healthy Participants (Part A), Participants With Active Systemic Lupus Erythematosus (Part B), and Healthy Participants of Chinese and Japanese Descent (Part C)
Brief Title: A Study of GSK4527363 in Healthy Participants, Systemic Lupus Erythematosus (SLE) Participants and Healthy Chinese and Japanese Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 221458
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Belimumab; First time in human study; GSK4527363; Healthy participants; Immunogenicity; Pharmacokinetics; Systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Part A: Healthy participants receiving GSK4527363 (Experimental)
  Interventions: Drug: GSK4527363
- Part A: Healthy participants receiving placebo matching GSK4527363 (Placebo Comparator)
  Interventions: Drug: Placebo matching GSK4527363
- Part A: Healthy participants receiving belimumab (Experimental)
  Interventions: Drug: Belimumab
- Part B: Participants with SLE receiving GSK4527363 (Experimental)
  Interventions: Drug: GSK4527363
- Part B: Participants with SLE receiving belimumab (Experimental)
  Interventions: Drug: Belimumab
- Part C: Healthy Japanese participants receiving GSK4527363 (Experimental)
  Interventions: Drug: GSK4527363
- Part C: Healthy Japanese participants receiving placebo matching GSK4527363 (Placebo Comparator)
  Interventions: Drug: Placebo matching GSK4527363
- Part C: Healthy Chinese participants receiving GSK4527363 (Experimental)
  Interventions: Drug: GSK4527363
- Part C: Healthy Chinese participants receiving placebo matching GSK4527363 (Placebo Comparator)
  Interventions: Drug: Placebo matching GSK4527363

INTERVENTIONS:
Drug: GSK4527363 — GSK4527363 will be administered to participants.
  Arms: Part A: Healthy participants receiving GSK4527363; Part B: Participants with SLE receiving GSK4527363; Part C: Healthy Chinese participants receiving GSK4527363; Part C: Healthy Japanese participants receiving GSK4527363
Drug: Placebo matching GSK4527363 — Placebo matching GSK4527363 will be administered to participants.
  Arms: Part A: Healthy participants receiving placebo matching GSK4527363; Part C: Healthy Chinese participants receiving placebo matching GSK4527363; Part C: Healthy Japanese participants receiving placebo matching GSK4527363
Drug: Belimumab — Belimumab will be administered to participants.
  Arms: Part A: Healthy participants receiving belimumab; Part B: Participants with SLE receiving belimumab

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of GSK4527363 in healthy participants (Part A), participants with active SLE (Part B), and healthy participants of Chinese and Japanese descent (Part C)

ELIGIBILITY:
Inclusion criteria:

For Part A and Part C (Healthy Participants):

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent form.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (vital signs and 12-lead ECG).
* Part C only: Be of Japanese (Cohort C1) or Chinese (Cohort C2) ancestry. i. Born in Japan (Cohort C1) or China mainland, Hong Kong or Taiwan (Cohort C2); and ii. Descendent of 2 ethnic Japanese (Cohort C1) or Chinese (Cohort C2) parents and 4 ethnic grandparents; and iii. Have lived outside Japan (Cohort C1) or China mainland, Hong Kong or Taiwan (Cohort C2) for less than 10 years at the time of screening.
* Body weight greater than or equals to (>=) 45 kilograms (kg).
* Body mass index (BMI) within the range 18-32 kilograms per square meter (kg/m^2) (inclusive).
* Male or female of non-childbearing potential

For Part B (SLE participants):

* 18 to 65 years of age inclusive, at the time of signing the informed consent form
* Documented clinical diagnosis of SLE according to the (European alliance of associations of rheumatology [EULAR]/ American College of Rheumatology [ACR] SLE classification criteria)
* Body weight >= 45 kg.
* BMI within the range 18-32 kg/m^2 (inclusive).
* Male or female

Exclusion criteria:

For Part A and Part C (Healthy Participants):

* History or presence or cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders.
* A history of recurrent infections, or treatment of a chronic infection within 3 months prior to the first dose of study drug.
* Any acute infection (including upper respiratory tract infections and urinary tract infections) which has not fully resolved within four weeks before dosing.
* Symptomatic herpes zoster within 3 months prior to screening.
* Have a history of malignancy, or a strong family history of malignancies related to immunosuppression.
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions.
* Abnormal blood pressure.
* Evidence of active or latent Tuberculosis (TB).
* Alanine transaminase (ALT) >=1.1* Upper limit of normal (ULN).
* Total bilirubin >1.0*ULN; Participants with Gilbert's syndrome can be included with total bilirubin >=1.5*ULN as long as direct bilirubin is <=1.5*ULN.
* Presence of Hepatitis B surface antigen (HBsAg) and Hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C Ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.
* Positive Human immunodeficiency virus (HIV) antibody test at screening.
* Prior medical history of anaphylaxis.
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 milliseconds (msec).
* Live vaccine(s) within 30 days before the dosing day or plans to receive such vaccines during the study.

For Part B (SLE participants):

* Any acute, severe lupus related flare during the Screening Period that needs immediate treatment.
* Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to SLE which, in the opinion of the principal investigator (PI), could confound the results of the clinical study or put the participant at undue risk.
* Have an acute or chronic infection requiring management as follows:

  i. Currently on any suppressive therapy for a chronic infection such as pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacteria.

ii. A serious infection requiring treatment with antibiotics and/or hospitalization if the last dose of antibiotics or the hospital discharge date was within 60 days of the first day of dosing (Day 1). Prophylactic anti-infective treatment is allowed.

* Evidence of active or latent TB.
* Confirmed Progressive Multifocal Leukoencephalopathy (PML) or unexplained new-onset or deteriorating neurologic signs and symptoms.
* ALT >2*ULN.
* Total bilirubin >1.5*ULN; Participants with Gilbert's syndrome can be included with total bilirubin >1.5*ULN as long as direct bilirubin is >1.5*ULN.
* Presence of HBsAg and/or HBcAb at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention.
* History or positive test at Screening for HIV.
* QTcF >450 msec.
* Solid or hematological malignancy or a history of malignancy (in the past 5 years) of except for basal cell or squamous cell in situ skin carcinomas, Cervical intraepithelial neoplasia (CIN) or carcinoma in situ of the cervix that have been resected with no evidence of metastatic disease for 3 years.
* Live or live-attenuated vaccine(s) within 30 days prior to Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2028-01-11 (Estimated); Study Completion 2028-01-11 (Estimated)

PRIMARY OUTCOMES:
Parts A, B and C: Number of participants with non-serious adverse events and serious adverse events | Up to Week 52
Parts A, B and C: Number of participants with clinically significant changes in physical examination, laboratory parameters, vital signs, and 12 lead electrocardiogram (ECG) findings | Up to Week 52
Parts A, B and C: Number of participants with clinically significant changes in Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Week 52
  The C-SSRS is an assessment tool that evaluates suicidal ideation and behavior. A suicidal ideation score will be calculated based on the maximum suicidal ideation category ranging from 1 to 5. Higher score indicates more suicidal ideation. A clinically important change in the C-SSRS is defined as a total score >0.

SECONDARY OUTCOMES:
Parts A and C: Area under the concentration-time curve to the last quantifiable concentration (AUC[0-t]) of GSK4527363 | Up to Week 52
Parts A and C: Area under the concentration-time curve to infinity (AUC[0-inf]) of GSK4527363 | Up to Week 52
Parts A and C: Maximum plasma concentration (Cmax) of GSK4527363 | Up to Week 52
Parts A and C: Apparent Terminal phase half-life (t1/2) of GSK4527363 | Up to Week 52
Parts A, B and C: Number of participants with anti-drug antibodies (ADAs) against GSK4527363 | Up to Week 52
Parts A, B and C: Titers of ADAs against GSK4527363 | Up to Week 52
Parts A, B and C: Percentage change from Baseline in cytokine levels | Baseline (Day 1) and up to Week 52
Part B: Area under the concentration-time curve to the end of the dosing period (AUC[0-tau]) of GSK4527363 | Up to Week 52
Part B: Maximum plasma concentration (Cmax) of GSK4527363 | Up to Week 52
Part B: Concentration at the end of the dosing interval (Ctrough) of GSK4527363 | Up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (3):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Columbus, Ohio
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Miguel de Tucumán
- Brazil (3):
  - GSK Investigational Site, Juiz de Fora
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Salvador
- Poland (4):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Sabadell Barcelona
  - GSK Investigational Site, Valladolid
- United Kingdom (3):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Middlesex

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/